CLINICAL TRIAL: NCT03523221
Title: Use of Dexamethasone in Prevention of the Second Phase or a Biphasic Reaction of Anaphylaxis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, DR. KHALID AL-ANSARI, Director of Pediatrics Emergency Centeres, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171661/17
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Anaphylaxis
Keywords: Mild -Moderate Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone arm (Active Comparator): All patients will be Urgently treated for anaphylaxis according to guideline protocol. Enrolled patients will be given one of study medication orally, and he /she will observe in the observation room with cardiac monitor and close monitoring by nurse.
  Interventions: Drug: Dexamethasone Oral
- Placebo arm (Placebo Comparator): All patients will be Urgently treated for anaphylaxis according to guideline protocol. Enrolled patients will be given one of study medication orally, and he /she will observe in the observation room with cardiac monitor and close monitoring by nurse.
  Interventions: Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Dexamethasone Oral — use of one dose of Dexamethasone orally.or placebo in addition to regular treatment of anaphylaxis

SUMMARY:
Anaphylaxis is an acute serious allergic reaction, with multi-organ system manifestations caused by the release of chemical mediators and it is potentially fatal .

Between 5% and 14% of patients may experience a recurrence of anaphylaxis 8-12 hours after the initial presentation, called biphasic (late-phase) .

The mainstay of treatment for children experiencing anaphylaxis remains adrenaline and H1-antihistamines. Corticosteroids are not life-saving and do not have an immediate effect on the symptoms of anaphylaxis but may help reduce or prevent a biphasic "late phase" reaction .

The aim of this study is to compare the efficacy of oral glucocorticoids in prevention of the second phase or biphasic reaction of anaphylaxis, as compared to placebo in children, presenting to the pediatric emergency department (PEC Al-Sadd) with mild to moderate anaphylaxis (Prospective Study).

Patients will be randomized to either one of the two treatment:

Treatment 1: Dexamethasone 0.6mg/kg oral. Treatment 2 : Placebo All patients will be urgently treated for anaphylaxis according to guideline protocol. Enrolled patients will be given one of the study medications orally, and he /she will observe in the observation room with cardiac monitor and close monitoring by nurse.

The treating physician will discharge patient when he/she looks well, breathing comfortably, has oxygen saturation >94%, stable blood pressure and no gastrointestinal or neurological manifestation.

Discharge patients will be sent home on anti-histamine (cetirizine) for 5days. All patients will be followed up for one week post discharge by a phone call asking about the general condition, relapse of symptoms, or need for readmission.

DETAILED DESCRIPTION:
Anaphylaxis is an acute serious allergic reaction, with multi-organ system manifestations caused by the release of chemical mediators . It requires immediate recognition and intervention.

The estimated rate of anaphylaxis in children was 10.5 per 100,000 persons-years . Although the Rochester Epidemiology Project showed a rate of 75.1 per 100,000 person-years in children aged 9 years and 65.2 per 100,000 person-years in children aged 10-19-years old.

In the state of Qatar with approximately 280,000 visits annually to Pediatric Emergency Center (PEC), there were 171 cases of anaphylaxis seen at the facility from September 2015 to September 2016.

Anaphylaxis is a clinical diagnosis based on typical systemic manifestations, due to exposure to a causative agent. There are many possible triggers, including food, medication, insect venoms, rubber latex and vaccines . In some individuals, anaphylaxis is idiopathic. Both IgE and non-IgE activation of mast cells and basophils that results in the release and production of several inflammatory and vasoactive substances, these substances most commonly involve the skin, respiratory, cardiovascular, and gastrointestinal systems. As a result, urticarial, angioedema, bronchospasm, laryngospasm, increased vascular permeability and decreased vascular tone.

Anaphylaxis involves a range of signs and symptoms from hives, wheezing and angioedema to cardiovascular collapse and death [9,10]. More than 80% of the patients will present with flushing, itching, hives, angioedema, or other skin or mucosal symptoms. Generally up to 70%, at least 2 organ systems (skin, respiratory, cardiovascular, gastrointestinal systems) are involved; however, only 10-45% have cardiovascular symptoms, including chest pain, hypotension, or shock . Between 5% and 14% of patients may experience a recurrence of anaphlactoid reaction 8-12 hours after the initial presentation, called Biphasic (late-phase) . Most of these reactions are mild or moderate . Risk factors for biphasic reactions include a severe initial reaction; presence of laryngeal edema or hypotension; delay in the administration of adrenaline (epinephrine); too small a dose of adrenaline; and a history of a previous biphasic reaction . Delayed symptoms can develop despite treatment .

The mainstay of treatment for children experiencing anaphylaxis remains adrenaline 1:1000 intramuscularly (IM) . H1-antihistamines are also commonly administered in anaphylaxis. The combination of H1 and H2 antihistamines appears to be more effective, especially for cutaneous symptoms . The onset of activity of these agents is slower than epinephrine and is considered next-in-line treatment.

International guidelines consider antihistamines and glucocorticoids as second-line . Corticosteroids are not life-saving and do not have an immediate effect on the symptoms of anaphylaxis, since it takes 4-6 hours to work.

Glucocorticoids are administered to 50% of individuals with anaphylaxis, despite a lack of compelling evidence supporting their use.

Recent retrospective study in emergency department, evaluated the association between glucocorticoids administration and prolonged length of stay. In 4years retrospective chart review study on anaphylaxis patient, 70% of study patients received glucocorticoids as part of their treatment. Glucocorticoids were not found to reduce follow up revisit in the three days post discharge. And it didn't decrease the likelihood of extra epinephrine need for flare of symptoms, and only found to decrease length of stay in severe anaphylaxis.

The existing evidence for the use of glucocorticoids appears to consist mainly of retrospective studies, case reports, and other descriptive literature. The need exists, however, for a prospective study on the use of glucocorticoids in the treatment of anaphylaxis and its effectiveness in prevention of biphasic reaction. The objective of the current study, therefore, is to complement the current research on anaphylaxis and to investigate if glucocorticoids are effective in the treatment of anaphylaxis and if it can prevent or limit biphasic reaction.

This will be the first randomized controlled trial to look at steroid use in anaphylaxis and its impact on anaphylaxis treatment on a prospective fashion which will be used to help standardize care in the use of steroid for this common condition.

ELIGIBILITY:
Inclusion Criteria:

* All patients 3 monthes-14years presenting to the Pediatric Emergency Department (AlSadd) with mild to moderate anaphylaxis

Exclusion Criteria:

Patients with severe anaphylaxis. Patient with history of immunological diseases. Patients on steroids therapy Patient with moderate-severe asthma on medication Patients with severe asthma

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Use of single dose of oral Dexamethasone decrease revisit to health center facility with relapse of anaphylaxis. | 2 years
  Would the use of single dose of oral Dexamethasone decrease revisit to health center facility with relapse of anaphylaxis signs and symptoms within one week after enrollment?

SECONDARY OUTCOMES:
use of oral Dexamethasone decrease the need for second dose of epinephrine after discharge from hospital. | 2 years
  Would the use of oral Dexamethasone decrease the need for second dose of epinephrine after discharge from hospital?

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Al ansari, FRCP, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al Sayyed R, Alansari K. Randomized blinded pilot trial of corticosteroid after mild-moderate anaphylaxis to prevent recurrence. Medicine (Baltimore). 2025 Aug 1;104(31):e43600. doi: 10.1097/MD.0000000000043600. PMID 40760578
- [Derived] Burroughs-Ray DC, Wells DR, Dennis MM, Jackson CD. Clinical Guideline Highlights for the Hospitalist: Anaphylaxis Management in Adults and Children. J Hosp Med. 2021 Feb;16(2):98-99. doi: 10.12788/jhm.3553. PMID 33496659